CLINICAL TRIAL: NCT04021420
Title: Safety and Efficacy of Blood Brain Barrier Opening With Implantable Device Sonocloud® Combined With Nivolumab Used Alone or an Association With Ipilimumab in Brain Metastases From Patients With Malignant Melanoma
Brief Title: Safety and Efficacy of Sonocloud Device Combined With Nivolumab in Brain Metastases From Patients With Melanoma
Acronym: SONIMEL01
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P160950J
Record Dates: First submitted 2019-07-01; First posted 2019-07-16 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Melanoma; Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- low intensity pulsed UltraSound (Experimental): SonoCloud® is an active implantable device (implantation duration until 16 weeks at maximum after inclusion). SonoCloud® delivers low intensity pulsed UltraSound (US). Along with systemic injection of an US resonator, SonoCloud® demonstrated safe and efficient at repetitively opening the BBB.
  Interventions: Device: SONOCLOUD; Drug: Nivolumab Injection

INTERVENTIONS:
Device: SONOCLOUD — The SonoCloud System is an active implantable medical. The SonoCloud is indicated to locally and transiently increase the permeability of the blood brain barrier to facilitate the passage of substances into the cerebral parenchyma.
  The SonoCloud System consists of :
  1. an implantable ultrasound transducer,
  2. a needle connection device,
  3. an external radiofrequency generator, and
  4. an ultrasound resonator. The SonoCloud® is designed to be fixed to the skull. The device is placed in a burr hole or in place of a bone flap and ultrasound energy is delivered directly to the brain tissue, without traversing the skull bone. The device is activated by connecting the implant to the external generator system using the transdermal needle. Once connected to the external generator, the implant delivers low-intensity pulsed UltraSound (US) for duration of 120-270 seconds. A total of 3 US dose levels will be evaluated (0.78, 0.9 and 1.03 MPa).
Drug: Nivolumab Injection — Nivolumab (flat dose: 240mg, 30 minutes infusion)

SUMMARY:
Anti PD-1 monoclonal antibodies (nivolumab and pembrolizumab) alone or in association with antiCTLA4 (Ipilimumab) are established as indisputable treatment of metastatic melanoma, with unprecedented overall survival, and are indicated for first-line treatment including patients with BRAF mutation. Given their high molecular weight, their penetration in the brain sanctuary is uncertain and relies on disruption of the Blood Brain Barrier (BBB) which occurs occasionally.

SonoCloud® is an implantable device delivering low intensity pulsed UltraSound (US). Along with systemic injection of an US resonator, SonoCloud® demonstrated safe and efficient at repetitively opening the BBB. The investigators anticipate that BBB opening could help at increasing brain penetration of monoclonal antibodies and potentially boosting immunity in the brain. This could translate in controlling brain disease with the same magnitude as for extra-cranial disease. This would also open avenues for optimizing the treatment of brain metastases in combination with checkpoint inhibitors in many other cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed metastatic melanoma
* Patients must have recovered from all side effects of their most recent systemic or local treatment for metastatic melanoma (grade ≤ 1).
* At least one measurable brain metastasis between 5 mm and 35 mm in diameter, not previously treated with surgery and/or radiosurgery and located less than 5 cm from the skull
* Patients may have received -or not- prior radiosurgery and/or surgery for brain metastases; if they have received prior local treatment, they must have at least 1new RANO and RECIST assessable brain metastases.
* BRAF status wild type or mutated (and in that case previous treatment with BRAF inhibitor and MEK inhibitor allowed)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1.
* Age >18 year
* Hemoglobin ≥10g/dl
* Platelets ≥ 100000mm3
* Neutrophils ≥1500/mm3
* Creatinine Clearance ≥ 50ml/mn
* AST <3N
* ALT<3N
* Total bilirubin <1.5N
* Alkaline phosphatase <3N
* INR < 1.5
* Prothrombin ≥70%
* TCA <1.2
* No Hepatocellular insufficiency
* No unhealed wound on the head
* No allergy to poly isoprene
* Signed informed consent
* Patient with health insurance coverage
* Life expectancy > 3 months

Exclusion Criteria:

* Patient previously treated by antiPD1 (except adjuvant antiPD1 therapy)
* Ocular melanoma
* Symptomatic or diffuse leptomeningeal involvement.
* Symptomatic hemorrhagic brain metastases.
* Symptoms of incoercible intracranial pressure; patients receiving corticosteroids and patients presenting intermittent seizures can be enrolled if they have a stable dose of corticosteroids (≤ 30mg/day corticotherapy) and anti-epileptic treatment since at least 2 weeks before enrolment.
* Indication for urgent neurosurgery or radiotherapy
* Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured or stage I untreated Chronic Lymphoid Leukemia.
* Known human immunodeficiency viruses (HIV) infection and any ongoing infectious disease or significant background.
* Concurrent administration of any anticancer therapies other than those administered in this study.
* Treatment with any cytotoxic and/or investigational drug, antiCTLA4 or targeted therapy ≤ 4 weeks or <5 half lives for targeted therapies or chemotherapy, prior to day 1 of study.
* Prior whole brain radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-07-05 (Estimated)

PRIMARY OUTCOMES:
Most Successful Dose (MSD) | Week 6
  Dose with the highest probability of BBB opening efficacy without toxicity directly related to the ultrasound emission.
  Toxicity evaluation:
  Safety will be assessed clinically and using brain Magnetic resonance imaging (MRI). An electroencephalogram will be performed only if clinically needed. Dose-Limiting-Toxicities (DLTs) evaluation will be done during the first 4 weeks of treatment for Nivolumab treatment and 6 weeks for Nivolumab + Ipilimumab treatment. DLTs directly related to the ultrasound emission are defined as occurrence of an adverse effect during the first administration of treatment, such as: :
  * neurological deficit within 2 days after the procedure and persistent at day 15;
  * localized brain edema not preexisting to the procedure;
  * occurrence of cerebral median line deviation not controlled by routine treatment or requiring salvage surgical procedure;
  * partial epilepsy induced or enhanced after the procedure and not control

SECONDARY OUTCOMES:
Best overall response rate, M3 | Month 3
  Best clinical objective response (BOR) (defined with the Response assessment in neuro-oncology criteria (RANO) and immunotherapy response assessment for neuro-oncology (iRANO) and the response evaluation criteria in solid tumours (RECIST) version 1.1 and the Immune-Related Response Criteria during the 3 first months
  RANO : Wen, Patrick Y., et al. "Updated response assessment criteria for high-grade gliomas: response assessment in neuro-oncology working group." J Clin Oncol 28.11 (2010): 1963-1972.
  iRANO : Okada, Hideho, et al. "Immunotherapy response assessment in neuro-oncology: a report of the RANO working group." The Lancet Oncology 16.15 (2015): e534-e542.
Overall response rate, M3 | Month 3
  Clinical objective response (defined with the RANO and iRANO and the RECIST version 1.1 and the Immune-Related Response Criteria) during the 3 first months
Best intracranial overall response rate (BICORR), M3 | Month 3
  Clinical efficacy will be assessed using TEP/TDM Scans (extracranial lesions) and MRI (intracranial metastases) at Month 3
Intracranial overall response rate (ICORR), M3 | Month 3
  Clinical efficacy will be assessed using TEP/TDM Scans (extracranial lesions) and MRI (intracranial metastases) at Month 3
Best extracranial overall response rate (BECORR), M3 | Month 3
  Best clinical objective response rate not taking account BICORR
Extracranial overall response rate (BECORR), M3 | Month 3
  Clinical objective response not taking account ICORR

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Louis Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided